CLINICAL TRIAL: NCT05023499
Title: Perioperative Glutamine Supplementation Restores Atrophy of Psoas Muscle in Gastric Adenocarcinoma Patients Undergoing Gastrectomy
Brief Title: Perioperative Glutamine Supplementation and Cachexia
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201909033RIND
Record Dates: First submitted 2021-08-15; First posted 2021-08-26 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Glutamine; Metabolic Disorder; Cachexia
Keywords: Gastric cancer; cachexia; psoas muscle; glutamine
MeSH Terms: conditions — Metabolic Diseases; Cachexia; Stomach Neoplasms | interventions — Powders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With glutamine supplementation: perioperative glutamine supplementation (PGS) was defined as the subjects with five-day parenteral plus one-month oral use.
  Interventions: Drug: SYMPT-X Glutamine, Oral Powder for Reconstitution
- Without glutamine supplementation: no glutamine use
  Interventions: Drug: SYMPT-X Glutamine, Oral Powder for Reconstitution

INTERVENTIONS:
Drug: SYMPT-X Glutamine, Oral Powder for Reconstitution — erioperative glutamine supplementation (PGS) was defined as the subjects with five-day parenteral plus one-month oral use.
  Other Names: SYMPT-X

SUMMARY:
Background Sarcopenia is characterized by the degenerative loss of skeletal muscle and is associated with increased adverse surgical outcomes. Glutamine is considered as an immune-modulating formula, which may stimulate protein synthesis in the skeletal muscle but also inhibited protein-degradation. In this study, the investigators calculate the area and volume psoas major muscle (PMMA; PMMV) of the third lumbar vertebral body as the reference of skeletal muscle. The aim of this study is to investigate whether perioperative glutamine supplementation restores atrophy of psoas muscle.

DETAILED DESCRIPTION:
A total of 550 gastric adenocarcinoma (GA) patients undergoing gastrectomy were enrolled for the study. Computed tomography was used to assess the short axis of the psoas muscle, and the change was calculated between preoperative day and three months after gastrectomy. Perioperative glutamine supplementation (PGS) was defined as the subjects with five-day parenteral plus one-month oral use. A linear regression model was performed to predict this association by adjusting clinic-demographics and nutritional calories.

ELIGIBILITY:
Inclusion Criteria:

* gastric cancer patients undergoing gastrectomy

Exclusion Criteria:

* hepatic or renal failures

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 550 gastric adenocarcinoma (GA) patients undergoing gastrectomy were enrolled for the study. Computed tomography was used to assess the short axis of the psoas muscle, and the change was calculated between preoperative day and three months after gastrectomy.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2021-08-14 (Actual)

PRIMARY OUTCOMES:
area psoas major muscle (PMMA; cm2) | 3 month after surgery
  We hypothesized that glutamine might play a role in improving sarcopenia. Both the PMMA and total volume of the psoas major muscle (PMMV) represent the severity of sarcopenia, because CT is routinely performed in surgical GA patients to check for cancer recurrence. The reason of including total volume into analysis is that it is considered a better index to define sarcopenia. [21] The primary and secondary endpoints were the perioperative change of PMMA and PMMV, respectively.
volume of psoas major muscle (PMMV; cm3) | 3 month after surgery
  We hypothesized that glutamine might play a role in improving sarcopenia. Both the PMMA and total volume of the psoas major muscle (PMMV) represent the severity of sarcopenia, because CT is routinely performed in surgical GA patients to check for cancer recurrence. The reason of including total volume into analysis is that it is considered a better index to define sarcopenia. [21] The primary and secondary endpoints were the perioperative change of PMMA and PMMV, respectively.

IPD SHARING:
Plan to Share IPD: No